CLINICAL TRIAL: NCT02539160
Title: Impact of Chronic Kidney Disease on the Pharmacodynamic and Pharmacokinetic Effects of Ticagrelor in Patients With Diabetes Mellitus and Coronary Artery Disease
Brief Title: Impact of Chronic Kidney Disease on the Effects of Ticagrelor in Patients With Diabetes and Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-10953
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Results first posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: coronary artery disease; diabetes mellitus; chronic kidney disease; ticagrelor
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Renal Insufficiency, Chronic | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CKD - Ticagrelor 90 (Active Comparator): Patients with chronic kidney disease will receive ticagrelor 90mg twice/daily for 7-10 days. Then patients will cross over to ticagrelor 60mg twice/daily for 7-10 days.
  Interventions: Drug: ticagrelor
- CKD - Ticagrelor 60 (Experimental): Patients with chronic kidney disease will receive ticagrelor 60mg twice/daily for 7-10 days. Then patients will cross over to ticagrelor 90mg twice/daily for 7-10 days.
  Interventions: Drug: ticagrelor
- Non-CKD - Ticagrelor 90 (Active Comparator): Patients without chronic kidney disease will receive ticagrelor 90mg twice/daily for 7-10 days. Then patients will cross over to ticagrelor 60mg twice/daily for 7-10 days.
  Interventions: Drug: ticagrelor
- Non-CKD - Ticagrelor 60 (Experimental): Patients without chronic kidney disease will receive ticagrelor 60mg twice/daily for 7-10 days. Then patients will cross over to ticagrelor 90mg twice/daily for 7-10 days.
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — Diabetic patients with or without chronic kidney disease will be randomized 1:1 to either (A) standard dose (90mg twice daily of ticagrelor) for 7-10 days and then cross-over to low dose (60mg twice daily of ticagrelor) for 7-10 days; (B) low dose (60mg twice daily of ticagrelor) for 7-10 days (phase 1) and then cross-over to standard dose (90mg twice daily of ticagrelor) for 7-10 days (phase 2).
  Other Names: brilinta

SUMMARY:
Patients with diabetes mellitus (DM) are at increased risk of atherothrombotic events. Importantly, DM is a key risk factor for the development of chronic kidney disease (CKD), which further enhances atherothrombotic risk. Clopidogrel is the most widely used platelet P2Y12 receptor inhibitor. However, despite its clinical benefit, patients with DM and CKD frequently experience recurrent atherothrombotic events. Ticagrelor is an oral, reversible, non-competitive P2Y12 receptor inhibitor with more potent and consistent platelet inhibition than clopidogrel. In large-scale clinical investigation, ticagrelor significantly reduced ischemic events to a greater extent than clopidogrel, a finding that was consistent also among DM patients. To date there has been no analysis on the efficacy of ticagrelor in DM patients according to CKD status. Moreover, although pharmacodynamic (PD) studies showed enhanced platelet inhibition associated with ticagrelor, it is unknown how this may be affected by CKD status. Ultimately, how PK/PD profiles of different ticagrelor dosing regimens may be affected by DM and CKD status is also unknown. The proposed study is aimed to show the impact of CKD status among patients with DM and coronary artery disease) CAD on PD and PK profiles of ticagrelor used at 2 doses (90mg bid and 60mg bid) in the setting of a prospective, randomized, cross-over trial.

DETAILED DESCRIPTION:
Patients with diabetes mellitus (DM) are at increased risk of atherothrombotic events. Importantly, DM is a key risk factor for the development of chronic kidney disease (CKD), which further enhances atherothrombotic risk. These observations underscore the importance of antiplatelet therapy for prevention of atherothrombotic recurrences in these high-risk patients. Clopidogrel is the most widely used platelet P2Y12 receptor inhibitor. However, despite its clinical benefit, patients with DM and CKD frequently experience recurrent atherothrombotic events. This may be in part due to the impaired pharmacokinetic (PK) and pharmacodynamic (PD) effects of clopidogrel in patients with DM and CKD. Since both DM and CKD represent pandemic public health problems, the prevalence of which will double over the next 20 years, identifying antiplatelet agents with more favorable PK/PD profiles is of key importance.

Ticagrelor is an oral, reversible, non-competitive P2Y12 receptor inhibitor with more potent and consistent platelet inhibition than clopidogrel. In large-scale clinical investigation, ticagrelor significantly reduced ischemic events to a greater extent than clopidogrel, a finding that was consistent also among DM patients. In patients with CKD, ticagrelor led to an even greater relative risk reduction of ischemic events, including cardiovascular mortality, compared to patients without CKD. However, to date there has been no analysis on the efficacy of ticagrelor in DM patients according to CKD status. Moreover, although PD studies showed enhanced platelet inhibition associated with ticagrelor, it is unknown how this may be affected by CKD status. Ultimately, how PK/PD profiles of different ticagrelor dosing regimens may be affected by DM and CKD status is also unknown. The proposed study is aimed to show the impact of CKD status among patients with DM and CAD on PD and PK profiles of ticagrelor used at 2 doses (90mg bid and 60mg bid) in the setting of a prospective, randomized, cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Type 2 DM, defined according to World Health Organization (WHO) definition, on treatment with oral hypoglycemic agents and/or insulin for at least 2 months without any changes in treatment regimen;
* Angiographically documented CAD.
* On treatment with low-dose aspirin (81mg/day) and clopidogrel (75mg/day) for at least 30 days as part of standard of care.

Exclusion Criteria:

* Patients with end-stage renal disease on hemodialysis.
* Use of any antiplatelet therapy (except aspirin and clopidogrel) in past 30 days.
* Use of parenteral or oral anticoagulation in past 30 day.
* Active pathological bleeding.
* History of intracranial hemorrhage with prior hemorrhage stroke.
* Blood dyscrasia or bleeding diathesis.
* Any active malignancy.
* Platelet count < 80x106/µl.
* Hemoglobin <10 g/dl.
* Known hepatic dysfunction (known moderate and severe hepatic dysfunction).
* Hemodynamic instability.
* Known allergy or hypersensitivity to ticagrelor or any excipients.
* Pregnant / lactating females (women of childbearing age must use reliable birth control while in the study).
* Strong inhibitors of cytochrome CYP3A4 and potent inducers of cytochrome CYP3A4 (to avoid interaction with ticagrelor): ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir and telithromycin.
* Patients with sick sinus syndrome (SSS) or high degree atrio-ventricular block without pacemaker protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Franchi F, Rollini F, Been L, Maaliki N, Abou Jaoude P, Rivas A, Zhou X, Jia S, Briceno M, Lee CH, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Bass TA, Angiolillo DJ. Impact of chronic kidney disease on the pharmacodynamic and pharmacokinetic effects of ticagrelor in patients with diabetes mellitus and coronary artery disease. Eur Heart J Cardiovasc Pharmacother. 2022 Aug 11;8(5):452-461. doi: 10.1093/ehjcvp/pvab042. PMID 34114623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between February 2016 and November 2019 at the outpatient clinics of University of Florida Health - Jacksonville (Jacksonville, Florida, USA).
Pre-assignment Details: 101 patients were consented and enrolled in the study; 9 patients were not eligible for randomization due to the presence of exclusion criteria. A total of 92 patients (non-CKD, n=48; CKD, n=44) were randomized and exposed to at least one dose of study medication.
Groups:
- DM-Non-CKD Ticagrelor 90 First: Patients with diabetes mellitus (DM) and coronary artery disease (CAD) were stratified according to chronic kidney disease (CKD) status. Non-CKD was defined by a glomerular filtrate rate (GFR) ≥ 60 ml/min/1.73m2.
  Non-CKD patients were randomized 1:1 to a) standard dose ticagrelor (90mg twice daily) for 7-10 days or b) low dose ticagrelor (60mg twice daily) for 7-10 days (phase 1). After 7-10 days of randomized treatment patients were crossed over to the alternative treatment, which was maintained for additional 7-10 days (phase 2).No wash out was performed.
- DM-Non-CKD Ticagrelor 60 First; DM-CKD Ticagrelor 90 First; DM-CKD Ticagrelor 60 First: Patients with diabetes mellitus (DM) and coronary artery disease (CAD) were stratified according to chronic kidney disease (CKD) status. CKD was defined by a glomerular filtrate rate (GFR) < 60 ml/min/1.73m2.
  CKD patients were randomized 1:1 to a) standard dose ticagrelor (90mg twice daily) for 7-10 days or b) low dose ticagrelor (60mg twice daily) for 7-10 days (phase 1). After 7-10 days of randomized treatment patients were crossed over to the alternative treatment, which was maintained for additional 7-10 days (phase 2). No wash out was performed.
Period: Phase 1 Pre-crossover
Arm/Group | DM-Non-CKD Ticagrelor 90 First | DM-Non-CKD Ticagrelor 60 First | DM-CKD Ticagrelor 90 First | DM-CKD Ticagrelor 60 First
Started | 24 | 24 | 22 | 22
Completed | 19 | 20 | 19 | 19
Not Completed | 5 | 4 | 3 | 3
Not completed — Adverse Event | 3 | 3 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Period: Phase 2 Post-crossover
Arm/Group | DM-Non-CKD Ticagrelor 90 First | DM-Non-CKD Ticagrelor 60 First | DM-CKD Ticagrelor 90 First | DM-CKD Ticagrelor 60 First
Started | 19 | 20 | 19 | 19
Completed | 19 | 20 | 19 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 77 patients (DM-CKD, n=38; DM-non-CKD, n=39) had pharmacodynamic (PD) data on study drug and represented the PD population that was used for the analysis.
Groups:
- DM-Non-CKD (All Participants Regardless of Sequence): Patients with diabetes mellitus (DM) and coronary artery disease (CAD) were stratified according to chronic kidney disease (CKD) status. Non-CKD was defined by a glomerular filtrate rate (GFR) ≥ 60 ml/min/1.73m2.
  Non-CKD patients were randomized 1:1 to a) standard dose ticagrelor (90mg twice daily) for 7-10 days or b) low dose ticagrelor (60mg twice daily) for 7-10 days (phase 1). After 7-10 days of randomized treatment patients were crossed over to the alternative treatment, which was maintained for additional 7-10 days (phase 2).
  This is a crossover study where participants in each cohort received both treatments but in difference sequences. Therefore, baseline characteristics are presented for the two separate cohorts but combining patients together regardless of treatment sequence.
- DM-CKD (All Participants Regardless of Sequence): Patients with diabetes mellitus (DM) and coronary artery disease (CAD) were stratified according to chronic kidney disease (CKD) status. CKD was defined by a glomerular filtrate rate (GFR) < 60 ml/min/1.73m2.
  CKD patients were randomized 1:1 to a) standard dose ticagrelor (90mg twice daily) for 7-10 days or b) low dose ticagrelor (60mg twice daily) for 7-10 days (phase 1). After 7-10 days of randomized treatment patients were crossed over to the alternative treatment, which was maintained for additional 7-10 days (phase 2).
  This is a crossover study where participants in each cohort received both treatments but in difference sequences. Therefore, baseline characteristics are presented for the two separate cohorts but combining patients together regardless of treatment sequence.
- Total: Total of all reporting groups
Arm/Group | DM-Non-CKD (All Participants Regardless of Sequence) | DM-CKD (All Participants Regardless of Sequence) | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 66 (9) | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 25 | 23 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 12 | 27
  White | 20 | 26 | 46
  More than one race | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
GFR [Mean (Standard Deviation); unit: ml/min/1.73m^2] | 88 (17) | 46 (9) | 67 (25)
Prior myocardial infarction [Count of Participants; unit: Participants] | 18 | 23 | 41

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured by Vasodilator Stimulated Phosphoprotein (VASP) Platelet Reactivity Index (PRI %)
Description: The primary end point of the study was platelet reactivity assessed by VASP-PRI following treatment with ticagrelor 90mg between DM-CKD and DM-non-CKD cohorts. PRI % is a measure of platelet reactivity, where higher PRI levels represent higher platelet reactivity and lower effect of antiplatelet medications. PRI greater than 50% represents inadequate response to antiplatelet medications.
Time Frame: 7 days
Population: The pharmacodynamic (PD) population included all patients with any PD data on study drug and without a major protocol deviation thought to affect significantly the PD findings. The PD population was used for analysis of all primary and secondary PD variables.
Measure: Mean (Standard Deviation); unit: PRI%
Arm/Group | CKD - Ticagrelor 90 | CKD - Ticagrelor 60 | Non-CKD - Ticagrelor 90 | Non-CKD - Ticagrelor 60
Number analyzed (Participants) | 38 | 38 | 39 | 39
PRI% | 25 (14) | 32 (13) | 31 (20) | 38 (20)
Statistical Analysis 1: Comparison: CKD - Ticagrelor 90 vs Non-CKD - Ticagrelor 90; Test type: Superiority; p = 0.105, t-test, 2 sided; Median Difference (Net) = 6.4, 95% CI 2-sided [-1.1 to 14.3]
Statistical Analysis 2: Comparison: CKD - Ticagrelor 60 vs Non-CKD - Ticagrelor 60; Test type: Superiority; p = 0.112, t-test, 2 sided; Mean Difference (Final Values) = 6, 95% CI 2-sided [-1.5 to 13.7]

2. Secondary Outcome: Platelet Reactivity Measured by VerifyNow P2Y12
Description: Platelet reactivity assessed by VerifyNow P2Y12 following treatment with ticagrelor 90mg or 60 mg between DM-CKD and DM-non-CKD cohorts. Results are expressed in P2Y12 reaction units (PRU). PRU is a measure of platelet reactivity, where higher PRU levels represent higher platelet reactivity and lower effect of antiplatelet medications. PRU greater than 208 represents inadequate response to antiplatelet medications.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: PRU
Arm/Group | CKD - Ticagrelor 90 | CKD - Ticagrelor 60 | Non-CKD - Ticagrelor 90 | Non-CKD - Ticagrelor 60
Number analyzed (Participants) | 38 | 38 | 39 | 39
PRU | 39 (57) | 59 (56) | 51 (52) | 74 (65)

ADVERSE EVENTS:
Time Frame: Any adverse event during the study period (any time from enrollment until completion of the study, up to 20 days) was recorded.
Arm/Group | CKD - Ticagrelor 90 | CKD - Ticagrelor 60 | Non-CKD - Ticagrelor 90 | Non-CKD - Ticagrelor 60
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/38 | 0/39 | 1/39
Other Adverse Events (participants affected / at risk) | 9/38 | 6/38 | 9/39 | 7/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CKD - Ticagrelor 90 (N=38) | CKD - Ticagrelor 60 (N=38) | Non-CKD - Ticagrelor 90 (N=39) | Non-CKD - Ticagrelor 60 (N=39)
hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypokalemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CKD - Ticagrelor 90 (N=38) | CKD - Ticagrelor 60 (N=38) | Non-CKD - Ticagrelor 90 (N=39) | Non-CKD - Ticagrelor 60 (N=39)
minor bleeding (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT02539160/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT02539160/ICF_001.pdf